CLINICAL TRIAL: NCT00873067
Title: Benefit of Complex Fractionated Atrial Electrograms Elimination in Atrial Fibrillation Ablation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fundacio Clinic Barcelona (Other)
Responsible Party: Principal Investigator, Josep Lluis Mont Girbau, Head of the Arrhythmia Unit, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCP/08/207-4495-CFAE
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2011-09

CONDITIONS: Atrial Fibrillation; Catheter Ablation
Keywords: Atrial fibrillation; Complex fractionated electrograms; CFAE
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACVP plus roof line (Active Comparator): Standard procedure for atrial fibrillation ablation, including pulmonary vein isolation plus roof line ablation. All ablation lines will be tested.
  Interventions: Procedure: Standard atrial fibrillation ablation procedure
- Additional CFAEs ablation (Active Comparator): Atrial fibrillation ablation with pulmonary vein ablation and roof line. In addition, complex fractionated atrial electrograms ablation will be performed, lasting at most 30 minutes.
  Interventions: Procedure: Additional Complex Fractionated Electrograms ablation

INTERVENTIONS:
Procedure: Additional Complex Fractionated Electrograms ablation — Atrial fibrillation ablation with pulmonary vein ablation and roof line. In addition, complex fractionated atrial electrograms ablation will be performed, lasting at most 30 minutes.
  Other Names: Complex atrial fractionated electrograms ablation
  Arms: Additional CFAEs ablation
Procedure: Standard atrial fibrillation ablation procedure — Standard procedure for persistent atrial fibrillation including circumferential pulmonary vein ablation and roof line, both being tested. No other lines or lesions will be performed.
  Other Names: ACVP ablation; Roof line
  Arms: ACVP plus roof line

SUMMARY:
The aim of this study is to evaluate whether performing complex fractionated atrial electrograms ablation improves outcomes in persistent or atrial fibrillation ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent (more than 7 days, or less than 7 days needing pharmacologic or electric cardioversion)
* Presence of atrial fibrillation at the beginning of the procedure

Exclusion Criteria:

* Hypo or hyperthyroidism
* Persistent long-lasting or non-defined duration atrial fibrillation
* Hypertrophic myocardiopathy
* Implantable defibrillation or pacemaker implanted
* Moderate or severe mitral valve disease or mitral prosthetic valve
* Ejection fraction less than 30%
* Left atrial anteroposterior diameter more than 50 mm.
* Previous atrial fibrillation ablation
* Contraindication to anticoagulation
* Left atrium thrombus
* Current infective disease or sepsis
* Pregnant women
* Current unstable angor
* Acute myocardial infarction in last 3 months
* Atrial fibrillation secondary to ionic disturbance, thyroids disease or secondary to any other reversible or non cardiovascular disease
* Reduced expectancy of life (less than 12 months)
* Patient participating in another clinical study that investigates a drug or device
* Psychologically unstable patient or denies to give informed consent
* Any cause that contraindicate ablation procedure or antiarrhythmic drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2009-01; Primary Completion 2012-02 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial arrhythmias without antiarrhythmic drugs | 1-year follow-up

SECONDARY OUTCOMES:
Freedom form atrial arrhythmias with or without antiarrhythmic drugs | 1-year follow-up
Presence of any complications in the acute phase or during follow-up | 1-year follow-up
Freedom from atypical atria flutter | 1-year follow-up
Increase in radioscopy time and radiofrequency application time | 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lluís Mont, MD, Study Chair — Hospital Clinic Universitary de Barcelona; Elena Arbelo, MD, PhD, Study Director — Hospital Clínic Universitari de Barcelona
Locations (1):
- Hospital Clinic Universitari de Barcelona, Barcelona, Barcelona, Spain